CLINICAL TRIAL: NCT04682678
Title: Spinal Cord Stimulation for Gait Disorders in Parkinson's Disease: a Pilot Study
Brief Title: Spinal Cord Stimulation for Gait Disorders in Parkinson's Disease
Acronym: SCM-PARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 38RC20.165; 2020-A02361-38 (Other: ID RCB)
Record Dates: First submitted 2020-12-08; First posted 2020-12-24 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OFF STIM (Sham Comparator): without stimulation
  Interventions: Procedure: Implantation of electrodes for Spinal cord stimulation
- ON STIM (Active Comparator): stimulation with the most effective parameters
  Interventions: Procedure: Implantation of electrodes for Spinal cord stimulation

INTERVENTIONS:
Procedure: Implantation of electrodes for Spinal cord stimulation — The implantation of electrodes for SCS at the epidural thoracic level connected to a neurostimulator at the abdominal level will be performed under general anaesthesia (hospitalization for 3 days in the Neurosurgery Department, CHUGA) in a maximum delay of 1 month following the preoperative assessment. During the first postoperative month, the optimization of SCS parameters will be performed by an experienced movement disorders neurologist.

SUMMARY:
Our project is based on the fundamental hypothesis that epidural spinal cord stimulation (SCS) improves Freezing of gait (FOG) in patients with Parkinson's disease. In eight patients implantation of electrodes for SCS at the epidural thoracic level will be performed under general anaesthesia.

Evaluation of gait and motor symptoms will be performed with and without stimulation, after a 3-month period for each of the stimulation conditions.This is a pilot, single centre, prospective, randomized, double blinded, cross-over study.

DETAILED DESCRIPTION:
Patients will be selected in the Movement Disorders Unit, Department of Neurology, University Hospital Grenoble. A preoperative assessment with gait assessment, clinical evaluation and Non-Motor Symptoms assessment will be realized. The implantation of electrodes for SCS at the epidural thoracic level connected to a neurostimulator at the abdominal level will be performed under general anaesthesia. During the first postoperative month, the optimization of SCS parameters will be performed by an experienced movement disorders neurologist.After the first post-operative month the patient will be randomized to the STIM ON condition (stimulation on, with the most effective parameters) or STIM OFF (without stimulation). The randomization will be performed in a double blinded fashion, by a neurologist working in open and not participating in the evaluations. After 3 months, the patient will be evaluated in a double blind condition, and the stimulation condition will be crossed for another period of 3 months. At the end of this second 3-month period, the patient will be again double-blind assessed. After this evaluation, the patient will enter the open phase of the study for a period of 6 months. For this last phase of the study, under STIM ON condition, an optimization of the stimulation settings will be realized, if necessary. At the end of this 6-month period of stimulation, the patient will be evaluated one last time. At all visits, clinical and gait evaluations will be carried out under chronic dopaminergic treatment. No change in antiparkinsonian treatment will be allowed during the entire study. Gait and clinical assessment will be performed at baseline and at the end of each double blinded phase and at 1-year follow-up. For the double-blind study the patient, the neurologist who performs the clinical evaluation and the expert who performs the gait test and analysis will be blind to the stimulation condition.

ELIGIBILITY:
Inclusion criteria:

1. Patients with diagnosis of idiopathic PD
2. Aged 50-85 years
3. Having a FOG (score> 14 at New-FOG-Questionnaire; score> = 1 at item 2.13 of the Movement Disorders Society-Unified Parkinson's Disease Rating Scale) despite the optimization of medical treatment
4. Drug treatment stable for at least 2 months
5. Able to give written consent.

Exclusion criteria:

1. Pain syndrome (score> = 2 at item 1.9 of the MDS-UPDRS II)
2. Psychosis
3. Severe depression
4. Severe cognitive impairment (Mini Mental Score Examination <19)
5. Patient receiving STN DBS treatment
6. Presence of other neurological or medical pathologies interfering with walking
7. Subject in period of exclusion from another study
8. Subject under administrative or judicial supervision
9. Subject who cannot be contacted in an emergency.
10. Person with any administrative or judicial measure of deprivation of rights and liberty

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
frequency and duration of Freezing Of Gait (FOG) episodes, objective | Month 6
  gait testing

SECONDARY OUTCOMES:
frequency and duration of Freezing Of Gait (FOG) episodes, subjective 1 | Month 12
  New FOG-questionnaire (NFOG-Q)
frequency and duration of Freezing Of Gait (FOG) episodes, subjective 2 | Month 12
  patient diary
impact of spinal cord stimulation on FOG, long term outcome | Month 12
  New Freezing Of Gait-questionnaire (NFOG-Q)
impact of spinal cord stimulation on quality of life, long term outcome | Month 12
  Parkinsons disease questionnaire (PDQ39)
impact of SCS on gait during a dual cognitive-motor task test | Month 12
  New FOG-questionnaire (NFOG-Q)
impact of SCS on other non-motor symptoms | Month 12
  SCales for Outcomes in PArkinson's disease - Autonomic Dysfunction (SCOPA-AUT)
impact of SCS on gait during timed up and go test | Month 12
  timed up and go test

CONTACTS AND LOCATIONS:
Overall Officials: Elena MORO, Principal Investigator — CHUGA
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No